CLINICAL TRIAL: NCT06752902
Title: Impact of a Personalised Prevention Approach on the Microbiological Homeostasis of the Oral Cavity During Fixed Orthodontic Treatment: Randomised Interventional Study
Brief Title: Personalised Prevention of Microbiological Homeostasis in the Oral Cavity During Fixed Orthodontic Treatment
Acronym: PREPERMIO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-AOI-04
Record Dates: First submitted 2024-10-11; First posted 2024-12-31 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Orthodontics
Keywords: oral dysbiosis; orthodontics; oral microbiotis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient with standard care (Other): patient with standard care
  Interventions: Other: Standard Care Arm
- patient with standard care combined with personalised prevention (Other): patient with standard care combined with personalised prevention
  Interventions: Other: standard care combined with personalised prevention

INTERVENTIONS:
Other: Standard Care Arm — standard care combined with personalised prevention
  Arms: patient with standard care
Other: standard care combined with personalised prevention — standard care combined with personalised prevention
  Arms: patient with standard care combined with personalised prevention

SUMMARY:
Oral dysbiosis systematically develops during orthodontic treatment [35][36]. Orthodontic appliances interfere with oral hygiene procedures and cause biofilm to accumulate, creating new retention zones, even in subjects who maintain correct oral hygiene [37]:

* A group benefiting from intensive personalised prevention
* A "conventionally monitored" group, with no personalised prevention. The hypothesis is that personalised prevention prevents dysbiosis from taking hold. If this hypothesis is confirmed, the concept could be extended to all patients, beyond orthodontics.

Based on the "biological signature" (microbiological and immune), a "risk profile" of patients could be defined, making it possible to better personalise the prevention message, the method applied and the frequency of follow-up. The aim would be to rebalance dysbiosis through a personalised prevention approach tailored to the profile defined.

It was decided to explore this hypothesis initially with orthodontic patients because they are "captive", i.e. in the course of treatment requiring regular visits. Prevention is aimed first and foremost at healthy patients, with the aim of maintaining them in good health. The project focuses on young patients undergoing orthodontic treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 to 20 (permanent dentition) requiring fixed orthodontic treatment.

Exclusion Criteria:

* Tobacco;
* Overcrowded restorations, untreated caries,
* lack of tooth mineralisation;
* Medical pathologies;
* Known immunodepression (congenital or acquired);
* Taking a treatment that may induce general immunodepression;
* Taking a probiotic;
* Taking a concomitant treatment that may interact with oral health

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-06-06 (Estimated)

PRIMARY OUTCOMES:
bacteria in biofilm | At inclusion
  number of pathogenic bacteria measured in the biofilm
bacteria in biofilm | At 3 months
  number of pathogenic bacteria measured in the biofilm
bacteria in biofilm | At 6 months
  number of pathogenic bacteria measured in the biofilm
bacteria in biofilm | At 9 months
  number of pathogenic bacteria measured in the biofilm
bacteria in biofilm | At 12 months
  number of pathogenic bacteria measured in the biofilm
viruses in biofilm | At inclusion
  number of viruses measured in the biofilm
viruses in biofilm | At 3 months
  number of viruses measured in the biofilm
viruses in biofilm | At 6 months
  number of viruses measured in the biofilm
viruses in biofilm | At 9 months
  number of viruses measured in the biofilm
viruses in biofilm | At 12 months
  number of viruses measured in the biofilm

SECONDARY OUTCOMES:
patient's satisfaction | at 12 months
  Patient satisfaction on a numerical scale from 0 to 10.
measurement of immune response | At inclusion
  assay of salivary cytokines in ng/ml
measurement of immune response | At 3 months
  assay of salivary cytokines in ng/ml
measurement of immune response | At 6 months
  assay of salivary cytokines in ng/ml
measurement of immune response | At 9 months
  assay of salivary cytokines in ng/ml
measurement of immune response | At 12 months
  assay of salivary cytokines in ng/ml
plaque index | through study completion, an average of 1 year
  scale QHI: quigley hein index
gingival index, | through study completion, an average of 1 year
  gingival index mesured with Ginigical Index Loe&Silness scale
toothbrush wear | through study completion, an average of 1 year
  toothbrush wear with the Toothbrush Wear Index (TWI)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Rance Orthodontics Practice, Dinan
  - Nice university hospital, Nice

IPD SHARING:
Plan to Share IPD: No